CLINICAL TRIAL: NCT07107711
Title: One-Stop Hybrid Versus Conventional Surgery for Acute Type A Aortic Dissection: A Randomized Controlled Trial
Brief Title: Hybrid vs. Conventional Surgery for Type A Aortic Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qi Hu, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020139
Record Dates: First submitted 2025-07-24; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Acute Stanford Type A Aortic Dissection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Hybrid Group (n=70) (Experimental): Patients were randomized to undergo one-stop hybrid surgery, which included total aortic arch replacement with a standard 4-branched artificial vascular graft combined with antegrade stent grafting of the proximal descending aorta, performed in a single stage under moderate hypothermia (approx. 28°C).
  Interventions: Procedure: One-Stop Hybrid Surgery
- Active Comparator: Conventional Group (n=70) (Active Comparator): Patients were randomized to undergo conventional total arch replacement using an integrated frozen elephant trunk (FET) hybrid prosthesis. The procedure was performed under deep hypothermic circulatory arrest (target temperature 23°C-25°C).
  Interventions: Procedure: Conventional Total Arch Replacement with Frozen Elephant Trunk

INTERVENTIONS:
Procedure: One-Stop Hybrid Surgery — With the patient under moderate hypothermia (approx. 28°C) and cardiopulmonary bypass, surgeons perform a total arch replacement using a standard 4-branched graft. After the open repair is complete, a separate, distinct covered stent graft is deployed antegradely into the descending aorta through the open distal end of the arch graft. Completion angiography confirms correct placement.
  Arms: Experimental: Hybrid Group (n=70)
Procedure: Conventional Total Arch Replacement with Frozen Elephant Trunk — With the patient under deep hypothermic circulatory arrest (23°C-25°C) and cardiopulmonary bypass, surgeons perform a total arch replacement using an integrated hybrid prosthesis (Frozen Elephant Trunk), which consists of a vascular graft sutured to a covered stent graft. This single device is deployed antegradely into the descending aorta, and the arch vessels are then reattached to the branches of the prosthetic graft.
  Arms: Active Comparator: Conventional Group (n=70)

SUMMARY:
This is a prospective, randomized controlled trial designed to compare the clinical efficacy and short-term outcomes of one-stop hybrid surgery versus conventional total arch replacement with frozen elephant trunk (FET) in patients with acute Stanford Type A Aortic Dissection. The study evaluates differences in perioperative metrics, postoperative complications, 30-day survival, aortic remodeling, and quality of life.

DETAILED DESCRIPTION:
Stanford Type A Aortic Dissection (TAAD) is a life-threatening condition requiring urgent surgical repair. This study tests the hypothesis that a one-stop hybrid surgery protocol is superior to conventional repair. 140 patients with acute TAAD were randomized to one of two groups. The experimental group received a one-stop hybrid surgery, which combines open total arch replacement using a standard branched surgical graft with the antegrade deployment of a separate stent graft, performed under moderate hypothermia. The active comparator group underwent conventional total arch replacement using an integrated frozen elephant trunk (FET) hybrid prosthesis, performed under deep hypothermic circulatory arrest. The study's main objective is to compare key clinical outcomes between the two surgical strategies, including a primary composite endpoint of 30-day mortality, stroke, and acute kidney injury, to provide evidence on the optimal surgical approach for this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years.
* Diagnosis of acute TAAD (symptom onset <72 hours) confirmed by imaging, with dissection involving the aortic arch requiring total arch replacement.
* Relative hemodynamic stability, defined as a systolic blood pressure >90 mmHg without high-dose vasopressor support (norepinephrine >0.1 µg/kg/min).
* Provision of informed consent.

Exclusion Criteria:

* Age >70 years.
* Stanford type B or non-dissection pathologies.
* Life-threatening comorbidities prohibitive of major cardiac surgery (e.g., advanced multiorgan failure from other causes, active malignancy).
* Absolute contraindications to surgery.
* History of previous ascending aorta or aortic arch surgery.
* Inability to provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence of the Composite Endpoint of 30-day Mortality, Stroke, and Acute Kidney Injury (Stage 2 or 3) | Within 30 days post-procedure
  A composite outcome measure including all-cause mortality, any new focal neurological deficit lasting >24 hours and confirmed by imaging (stroke), and acute kidney injury defined as Stage 2 or 3 by KDIGO criteria. The measure is the percentage of patients in each group who experience at least one of these events.

SECONDARY OUTCOMES:
All-Cause Mortality at 30 Days | Within 30 days post-procedure
  The percentage of patients who died from any cause.
Incidence of Postoperative Stroke | Within 30 days post-procedure
  The percentage of patients with a new focal neurological deficit lasting >24 hours, confirmed by imaging.
Incidence of Stage ≥2 Acute Kidney Injury (AKI) | Within 30 days post-procedure
  The percentage of patients developing AKI Stage 2 or 3, as defined by KDIGO criteria.
Operative Metrics | Intraoperative
  Includes total operative time, cardiopulmonary bypass duration, and aortic cross-clamp duration. Measured in minutes or hours.
Duration of Mechanical Ventilation | During the postoperative hospital stay (up to 30 days post-procedure)
  The total time a patient requires mechanical ventilation support after surgery, measured in hours.
Incidence of Other Major Postoperative Complications | During hospital stay (up to 30 days post-procedure)
  Includes pulmonary infection, severe hypoxemia, postoperative delirium (assessed via CAM-ICU), and reoperation for bleeding.
Change in Aortic Morphology Score | 1 Month Post-procedure, 3 Months Post-procedure
  Aortic remodeling assessed by a 7-parameter scoring system on Magnetic Resonance Imaging (MRI). The score ranges from 0 to 16, with lower scores indicating more favorable remodeling (a better outcome).
Change in Quality of Life | 3 Months Post-procedure
  Assessed using the Kansas City Cardiomyopathy Questionnaire (KCCQ) summary score. The score ranges from 0 to 100, where higher scores indicate better quality of life (a better outcome).
Incidence of Endoleak | 1 Month Post-procedure, 3 Months Post-procedure
  Presence of any endoleak detected on follow-up MRI.
Incidence of Cardiovascular Events | Through study completion (3 months)
  Number of patients experiencing major adverse cardiovascular events (e.g., myocardial infarction, repeat aortic intervention) during follow-up.
Length of Intensive Care Unit (ICU) Stay | During the postoperative hospital stay (up to 30 days post-procedure)
  The total number of days a patient stays in the Intensive Care Unit (ICU) following surgery.
Total Postoperative Hospital Stay | During the postoperative hospital stay (up to 30 days post-procedure)
  The total number of days from surgery until hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China